CLINICAL TRIAL: NCT05828784
Title: Italian Title:STUDIO CLINICO LONGITUDINALE, PROSPETTICO, PRE-CE PER LA VALUTAZIONE DELLA EFFICACIA E DELLA SICUREZZA DI UN CAGE INTERVERTEBRALE IN TITANIO ASSOCIATO AD UN SOSTITUTO OSSEO SINTETICO DI NATURA BIOCERAMICA NELLA NORMALE PRASSI CLINICA IN PROCEDURE DI FUSIONE INTERVERTEBRALE English Title: LONGITUDINAL, PROSPECTIVE, PRE-CE CLINICAL STUDY TO EVALUATE THE EFFICACY AND SAFETY OF A TITANIUM INTERVERTEBRAL CAGE ASSOCIATED WITH A BIOCERAMIC SYNTHETIC BONE SUBSTITUTE IN NORMAL CLINICAL PRACTICE IN INTERVERTEBRAL FUSION PROCEDURES
Brief Title: SPACE (SPS ADVANCED CAGE): SPS Spacer for Intervertebral Fusion, Longitudinal, Prospective Clinical Study
Acronym: SPACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SPS srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPS101
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Treatment of Degenerative Diseases of the Spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 35 consecutive patients (Other)
  Interventions: Device: Intersomatic arthrodesis

INTERVENTIONS:
Device: Intersomatic arthrodesis — Arthrodesis is an operative modality also used in the treatment of multiple recurrences of herniated discs, stenosis (narrowing) of the spinal anal, degenerative and malformative spondylolisthesis.
  The procedure can be performed with different surgical techniques, but in all cases it aims to achieve the same goal: to re-establish, through the use of spacers, the correct distance between two vertebral somes, in cases of disc degeneration, that are no longer able to fulfill their function; that is, they no longer absorb mechanical stresses and/or compress the nerve structures of the spine causing almost always unbearable (disabling) pain.

SUMMARY:
Space clinical study aims to evaluate the performance, in terms of efficacy and safety of an intervertebral spacer associated with a bioceramic bone substitute in the context of intervertebral surgery for degenerative diseases.

Specifically, it is intended to evaluate:

* the capacity for bone regeneration/fusion, defined as absence of loosening and presence of continuous trabecular bone bridge in the absence of radiolucency lines, verified by imaging (CT) and evaluated according to the Brantingan scale;
* the safety of the medical device, through the incidence of any adverse events, complications, unexpected reactions, accidents;
* the improvement of clinical outcome in terms of pain and disability, at 9/14 months follow-up compared with preoperative scores, by clinical indices such as ODI and VAS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided hospital consent for surgical treatment;
* Male patients and non-pregnant female patients between the ages of 18 and 75 years;
* Patients requiring single-level interbody fusion in the L3-L4 and L4-L5 tract;
* Patients with degenerative diseases of the spine, such as lumbar canal stenosis, lumbar discopathy, degenerative spondylolisthesis grade I;
* Patients with a BMI <= 30;
* Patients physically and mentally willing and able to comply with postoperative indications;
* Patient able to understand the Italian language;
* If the investigator decides to fuse an additional level for spinal stability during surgery, this is not an exclusion criterion; however, only one level will be measured to comply with the surgical indication.
* Female patients who are pregnant or planning to become pregnant during the course of the study;
* Obese patients with a BMI index > 30.

Exclusion Criteria:

Patients with:

* systemic or localized infection;
* Inflammatory or autoimmune disease;
* hypercalcemia;
* coagulation disorders;
* metabolic disorders;
* insulin-dependent diabetes;
* alterations or complications of thyroid function;
* overt allergy to calcium phosphate salts;
* self-reported allergies to drugs and/or medical devices;
* tumor and/or infectious diseases of the spine;
* active neoplasms;

In addition, patients who:

* Abuse alcohol and drugs;
* Are affected by smoking (> 20 cigarettes/day);
* Are on drug therapy that causes alteration of bone regeneration (e.g., chemotherapy);
* already had surgery (revision surgery).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Bone fusion rate | 9 months
  the evaluation of the success rate in achieving bone fusion defined as bone regeneration/fusion capacity, understood as lack of loosening and presence of continuous trabecular bone bridge in the absence of radiolucency lines, verified by diagnostic imaging (CT) and evaluated according to the Brantingan scale;

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria, Italy